CLINICAL TRIAL: NCT05411770
Title: Investigation of The Relationship Between The Stomatognathic System, Spine Posture and Pelvic Symmetry in Adolescence Individuals
Brief Title: The Relationship Between The Stomatognathic System, Spine Posture And Pelvic Symmetry
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/09
Record Dates: First submitted 2022-05-31; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Stomatognathic System; Spine; Pelvis; Posture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Thoracic kyphosis and lumbar lordosis angle assessment — Thoracic kyphosis and lumbar lordosis angle assessment was performed with the reliable Baseline Bubble Inclinometer®.
Device: Temporomandibular range of motion — TMJ range of motion, maximum mouth opening amount (MAAM), right and left lateral movements of the mandible (laterotrusion), anterior movement of the mandible (protrusion), and backward movement of the mandible (retrusion) were measured with a millimetric ruler, while the adolescent was seated on a chair.
Device: Measuring the cervical joint range of motion — Cervical joint flexion, extension, lateral flexion and rotation ranges of motion were measured with a universal goniometer while the adolescent was sitting in a chair.
Device: Craniovertebral angle measurement — Head posture of the adolescent was evaluated by craniovertebral angle (CVA) method. Adolescents sat on a chair with back support in an upright position and turned sideways to the worker. The pivot point was accepted as the seventh cervical vertebra, and the angle between the head (tragus) and the horizontal plane was measured with a goniometer and recorded in degrees.
Device: Tragus-to-wall distance measurement — Tragus-to-wall distance was measured using a tape measure and recorded in cm.
Device: Scoliosis angle assessment — Scoliosis angle assessment was done with a scoliometer.

SUMMARY:
This study was planned to examine the relationship between the stomatognathic system, spine posture and pelvis symmetry. 91 healthy adolescence were included in the study. For stomatognathic system, temporomandibular range of motion with millimeter ruler, cervical joint range of motion and craniovertebral angle measurement with goniometer, tragus-wall distance measurement with tape measure, kyphosis and lordosis angle measurement with Baseline Bubble Inclinometer®, trunk rotation angle scoliometer for scoliosis, lower extremity length measurements for pelvis symmetry were made using a tape measure.

ELIGIBILITY:
Inclusion Criteria:

* No known neurological, rheumatological, musculoskeletal problems
* Has no visual or hearing impairment
* Ability to adapt to the parameters to be applied in the study
* Ability to perform tests to be applied
* Consists of voluntary adolescent individuals whose families gave permission to participate in the study.

Exclusion Criteria:

* Receiving joint sounds in the form of clicks or crepitations from the TMJ during mouth opening and closing or chewing
* Passion and tenderness in the TMJ on palpation
* Having a tumor Having received orthodontic treatment in the last 3 years
* Having a history of head, neck and maxillofacial surgery

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Healthy adolescent individuals aged 10-18 years were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Thoracic kyphosis and lumbar lordosis angle assessment | 12 Weeks
  Thoracic kyphosis and lumbar lordosis angle assessment was performed with the reliable Baseline Bubble Inclinometer®.
Temporomandibular range of motion | 12 Weeks
  TMJ range of motion, maximum mouth opening amount (MAAM), right and left lateral movements of the mandible (laterotrusion), anterior movement of the mandible (protrusion), and backward movement of the mandible (retrusion) were measured with a millimetric ruler, while the adolescent was seated on a chair and recorded in mm.
Measuring the cervical joint range of motion | 12 Weeks
  Cervical joint flexion, extension, lateral flexion and rotation ranges of motion were measured with a universal goniometer while the adolescent was sitting in a chair.
Craniovertebral angle measurement | 12 Weeks
  Head posture of the adolescent was evaluated by craniovertebral angle (CVA) method. Adolescents sat on a chair with back support in an upright position and turned sideways to the worker. The pivot point was accepted as the seventh cervical vertebra, and the angle between the head (tragus) and the horizontal plane was measured with a goniometer and recorded in degrees.
Tragus-to-wall distance measurement | 12 Weeks
  Tragus-to-wall distance was measured using a tape measure and recorded in cm.
Scoliosis angle assessment | 12 Weeks
  Scoliosis angle assessment was done with a scoliometer.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Betül Demirkapi, MSc, Principal Investigator — Sanko University
Locations (1):
- Sanko University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No